CLINICAL TRIAL: NCT00169559
Title: A Multi-center, Three-staged, Randomized, Parallel Group, Sequential, Double-blind, fenofibrate-and Placebo-controlled Dose-response Evaluation of the Safety, Tolerability, and Effects on Plasma HDLc and TG of Eight Weeks Treatment With 1µg to 20µg Daily Doses of GW590735 in Otherwise Healthy Subjects With Low HDLc, Mildly to Moderately Elevated TG, and Normal LDLc
Brief Title: Dyslipidemia Study Investigating The Increase In "Good Cholesterol"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAA20001
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Dyslipidaemias
Keywords: triglycerides; Hypertriglyceridemia; cholesterol; LDL; HDL
MeSH Terms: conditions — Hypertriglyceridemia | interventions — 2-methyl-2-(4-(((4-methyl-2-(4-trifluoromethylphenyl)-thiazol-5-ylcarbonyl)amino)methyl)phenoxy)propionic acid; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Placebo Comparator): Placebo
  Interventions: Drug: GW590735; Drug: fenofibrate
- Arm 2 (Active Comparator): Fenofibrate
  Interventions: Drug: GW590735

INTERVENTIONS:
Drug: GW590735 — 1µg to 20µg daily doses of GW590735
Drug: fenofibrate — Marketed Drug
  Arms: Arm 1

SUMMARY:
An eight week comparison of the investigational drug GW590735, placebo, and the marketed drug fenofibrate intended to increase the levels of "good cholesterol" and decrease levels of "bad cholesterol" in healthy patients with low levels of good cholesterol and high levels of bad cholesterol.

DETAILED DESCRIPTION:
A multi-center, three-staged, randomized, parallel group, sequential, double-blind, fenofibrate-and placebo-controlled dose-response evaluation of the safety, tolerability, and effects on plasma HDLc and TG of eight weeks treatment with 1µg to 20µg daily doses of GW590735 in otherwise healthy subjects with low HDLc, mildly to moderately elevated TG, and normal LDLc

ELIGIBILITY:
Inclusion criteria:

* High-density lipoprotein cholesterol less than or equal to 45 mg/dL.
* Triglycerides greater than or equal to 120 mg/dL and less than or equal to 500 mg/dL.
* Women must be surgically sterile or postmenopausal.

Exclusion criteria:

* Heart disease
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-11; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
change from baseline in fasting plasma HDLc concentration at the end of eight weeks of double blind treatment | 8 weeks

SECONDARY OUTCOMES:
changes from baseline in: fasting plasma total cholesterol, TG, LDLc, ApoA1, ApoA2, Lipoprotein containing ApoA1 and not ApoA2, Lipoprotein containing both ApoA1 and ApoA2, Apo B100, Apo CIII, Free Fatty Acid, insulin, fibrinogen, and C-reactive protein | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (41):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Healdsburg, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Lauderale, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Orland Park, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Conroe, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec